CLINICAL TRIAL: NCT07278284
Title: The Effectiveness of Press Needle Acupuncture on Preoperative Anxiety in Tympanoplasty and Mastoidectomy at RSUD Kabupaten Tangerang
Brief Title: The Effectiveness of Press Needle Acupuncture on Preoperative Anxiety in Tympanoplasty and Mastoidectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Miranda Hartini Marpaung, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-11-1709
Record Dates: First submitted 2025-11-26; First posted 2025-12-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The press needle acupuncture therapy will be designated as the intervention group, while the sham press needle acupuncture therapy will be designated as the control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Press Needle Acupuncture
  Interventions: Device: The press needle acupuncture
- Control Group (Sham Comparator): Sham press needle acupuncture
  Interventions: Device: The sham press needle acupuncture

INTERVENTIONS:
Device: The press needle acupuncture — Insertion of acupuncture needles (Pyonex, Korea) measuring 0.2 × 0.9 mm at the auricular acupuncture points Micro Acupuncture - Triangular Fossa1 (MA-TF1) Shenmen, Micro Acupuncture - Anti Tragus2 (MA-AT2) Thalamus, and Micro Acupuncture - Inferior Concha7 (MA-IC7) Heart unilaterally (on the ear opposite to the surgical side), and insertion of a 0.2 × 1.5 mm press needle at the body point Extra - Head Neck3 (EX-HN3). The needles are inserted one day before surgery, with no stimulation performed either during insertion or while the press needles remain in place. Participants are instructed not to touch the application sites until the needles are removed.
  Arms: Intervention Group
Device: The sham press needle acupuncture — Application of round adhesive patches with a diameter resembling that of a press needle at the auricular points Micro Acupuncture - Triangular Fossa1 (MA-TF1) Shenmen, Micro Acupuncture - Anti Tragus2 (MA-AT2) Thalamus, and Micro Acupuncture - Inferior Concha7 (MA-IC7) Heart unilaterally (on the ear opposite to the surgical side), as well as at the body point Extra - Head Neck3 (EX-HN3). The patches are applied one day before surgery, with no stimulation performed either during application or while the patches remain in place. Participants are instructed not to touch the application sites until the patches are removed.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if press needle acupuncture works to treat preoperative anxiety in Tympanoplasty and Mastoidectomy at RSUD Kabupaten Tangerang in adults. The main questions it aims to answer are:

Does the press-needle acupuncture administered one day before tympanoplasty and mastoidectomy significantly reduce preoperative anxiety levels-measured using the Amsterdam Preoperative Anxiety and Information Scale (APAIS)-compared with the sham press-needle group at 30 minutes after the intervention and 60 minutes before anesthesia induction?

Is there a difference in effectiveness between press-needle acupuncture and sham press-needle acupuncture in influencing Heart Rate Variability (HRV) among patients undergoing tympanoplasty and mastoidectomy at 30 minutes after the intervention, 60 minutes before anesthesia induction, 2 hours postoperatively, and 24 hours postoperatively?

Are there any adverse events associated with the use of press-needle acupuncture and sham press-needle acupuncture in patients with preoperative anxiety undergoing tympanoplasty and mastoidectomy?

Participants will:

Receive press-needle acupuncture or sham press-needle acupuncture one day before surgery Have the press needles left in place for a total of 3 days Undergo removal of the needles before hospital discharge Complete preoperative anxiety assessments and routine monitoring according to the study schedule

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed and scheduled for elective tympanoplasty and mastoidectomy under general anesthesia who experience preoperative anxiety.
* Patients aged 18-59 years.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Patients who have not taken any anti-anxiety medication within the past 24 hours.
* Willing to participate in the study until completion and sign the informed consent form.

Exclusion Criteria:

* Patients with a history of psychiatric disorders or those taking psychotropic medications.
* Presence of contraindications to acupuncture, including medical emergencies, pregnancy, thrombocytopenia with platelet count <50,000/µL, and any history of bleeding disorders.
* Presence of infection, scarring, or malignancy at the acupuncture site.
* Anatomical abnormalities of the auricle.
* History of hypersensitivity reactions to prior acupuncture therapy (such as metal allergy, keloids, or other cutaneous hypersensitivity reactions).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Baseline, 30 minutes post-intervention, 60 minutes before anesthesia induction
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a questionnaire consisting of six items rated on a 5-point Likert scale. These six items are divided into three components: anxiety related to anesthesia, anxiety related to the surgical procedure, and the need-for-information component. Higher scores indicate higher levels of preoperative anxiety and a greater need for information.
Heart Rate Variability (HRV) | Baseline, 30 minutes post-intervention, 60 minutes before anesthesia induction, 2 hours postoperatively, 24 hours postoperatively
  Heart rate variability measurements using an HRV monitor (Polar H10) for 5 minutes in the seated position, with the corresponding application operated on the research assistant's smartphone.

SECONDARY OUTCOMES:
Side effects | Immediately after the intervention
  Reactions that occur during or after press-needle application, documented observationally using a monitoring sheet.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — the Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No